CLINICAL TRIAL: NCT01722253
Title: Postoperative Analgesia After Low Frequency Electroacupuncture as Adjunctive Therapy in Inguinal Hernia Surgery With Abdominal Wall Mesh Reconstruction
Brief Title: Postoperative Analgesia After Low Frequency Electroacupuncture
Acronym: LFE
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Maria I. Dalamagka, consultant Anaesthesiologist, Aristotle University Of Thessaloniki
Other Study IDs: 225
Record Dates: First submitted 2012-11-03; First posted 2012-11-06 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Inguinal Hernia
Keywords: electroacupuncture; acupuncture; pain management
MeSH Terms: conditions — Hernia, Inguinal; Agnosia | interventions — Electroacupuncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- placebo, electroacupuncture: Electroacupuncture before and after surgery (40min and 60 min respectively) with frequency 2 Hz, and 'frequency scanning mode'.
  Placebo electroacupuncture, in which the needles are secured (without penetrating the skin) and connected to the electrical device, which is not functional.
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — Electrical stimulation device with frequency 2 Hz and 'frequency scanning mode'

SUMMARY:
The purpose of this study is to determine whether electroacupuncture is a effective tool to the postoperative analgesia

DETAILED DESCRIPTION:
The electroacupuncture is a known therapeutic modality with particular application to pain. In this study the investigators investigate the effect of electroacupuncture in condition of surgery, which is a particularly painful situation. The investigators will verify the postoperative analgesia, as patients will receive either electroacupuncture or placebo electroacupuncture.

ELIGIBILITY:
inclusion criteria:

* healthy male volunteers
* 18-75 years old

Exclusion Criteria:

* bilateral or recurrent hernia
* significant cardiovascular, pulmonary, renal, hepatic, neurological disease
* psychiatric history
* use of opioids until the last month
* body mass index greater than 30
* treatment with beta-blockers
* aged over 75
* previous experience with acupuncture
* hypersensitivity to opioids
* pacemaker patient
* patients being treated with monoamine oxidase inhibitors and selective serotonin reuptake inhibitors.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the Surgical Clinic with right or left inguinal hernia, residents of Thessaly, Greece.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2008-12; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Monitoring of pain with the Visual Analogue scale within the first 24 hours after surgery | within the first 24 hours after surgery
  Monitoring of pain with the Visual Analogue scale performed preoperatively and at 30, 90 min, 10 hours and 24 hours after surgery

SECONDARY OUTCOMES:
Control of anxiety with the State-Trait Anxiety Inventory within 24 hours after surgery | within the first 24 hours after surgery
  The State-Trait Anxiety Inventory performed preoperatively and at 30, 90 min, 10 hours and 24 hours after surgery

OTHER OUTCOMES:
Monitoring of pain with the use of an algometer within the first 24 hours after surgery | within the first 24 hours after surgery
  Monitoring of pain with the use of an algometer performed preoperatively and at 30, 90 min, 10 hours and 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios G Vasilakos, Professor, Study Chair — Aristotle University; Maria I Dalamagka, consultant, Principal Investigator — Aristotle University
Locations (1):
- Aristotle University, Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Derived] Dalamagka M, Mavrommatis C, Grosomanidis V, Karakoulas K, Vasilakos D. Postoperative analgesia after low-frequency electroacupuncture as adjunctive treatment in inguinal hernia surgery with abdominal wall mesh reconstruction. Acupunct Med. 2015 Oct;33(5):360-7. doi: 10.1136/acupmed-2014-010689. Epub 2015 Jun 3. PMID 26040491